CLINICAL TRIAL: NCT00218218
Title: Transdermal Nicotine and Bupropion for Smoking in Schizophrenics (Study 1)
Brief Title: Effects of Transdermal Nicotine on Smoking, Craving and Withdrawal in People With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jennifer W. Tidey, Brown University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NIDA-14002-1; R01-14002-1; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Tobacco Use Disorder; Schizophrenia
Keywords: Nicotine Dependence; Tobacco Dependence
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Tobacco Use Disorder; Schizophrenia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Transdermal nicotine, 42 mg
  Interventions: Drug: Transdermal Nicotine Patch
- 2 (Experimental): Transdermal nicotine, 21 mg
  Interventions: Drug: 21 mg transdermal nicotine
- 3 (Placebo Comparator): placebo patch
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: Transdermal Nicotine Patch — 42 mg transdermal nicotine
  Other Names: nicotine patch
  Arms: 1
Drug: 21 mg transdermal nicotine
  Other Names: nicotine patch
  Arms: 2
Drug: placebo patch
  Arms: 3

SUMMARY:
Individuals with schizophrenia are three times as likely to smoke cigarettes as individuals without schizophrenia. While a great deal of research has been focused on smoking cessation programs for healthy individuals, little attention has been directed towards developing an effective smoking cessation treatment for schizophrenics. This project will evaluate the effects of 0, 21 and 42 mg transdermal nicotine on smoking, urge to smoke, and nicotine withdrawal symptoms after 5 hrs abstinence in smokers with schizophrenia and heavy-smoking non-psychiatric control smokers.

DETAILED DESCRIPTION:
Nicotine is the most commonly abused drug among individuals with schizophrenia; at least 60 percent of schizophrenics smoke cigarettes. Nicotine withdrawal may cause a temporary worsening of schizophrenia symptoms, making it especially difficult for these individuals to quit smoking. Little research has been done on the most effective way to control nicotine use in schizophrenic individuals. Transdermal nicotine and bupropion reduce smoking in non-psychiatric smokers, but little is known about the effects of these medications in smokers with schizophrenia. This project examines the effects of 0, 21 and 42 mg transdermal nicotine on smoking behavior and related subjective effects (urge to smoke and nicotine withdrawal symptoms) in smokers with schizophrenia and non-psychiatric heavy smoking controls. Participants come to the laboratory at 9 am, at which time placebo or nicotine patches are applied. After 5 hrs of smoking abstinence, participants undergo a smoking cue reactivity assessment in which craving and withdrawal symptoms are measured after viewing and handling neutral cues and smoking cues. This is followed by 90 min period in which participants can smoke freely, and smoking topography variables are measured.

ELIGIBILITY:
Inclusion Criteria:

* Smokes between 20 and 50 cigarettes per day
* Diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* If enrolled in the control group, must not be diagnosed with a psychiatric disorder
* Currently dependent on alcohol or any drug (other than nicotine)
* Currently trying to quit smoking
* Currently taking bupropion, desipramine, clonidine, buspirone, or doxepin
* History of liver disease
* History of heart attacks or chest pain
* Allergic to adhesives
* Pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-06; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Smoking behavior (measured by automated topography) | after 5 hrs abstinence

SECONDARY OUTCOMES:
Adverse events (measured by self-report throughout the study) | ongoing
Nicotine withdrawal severity | after 5 hrs abstinence
Smoking urge | after 5 hrs withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer W. Tidey, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Providence VA Medical Center, Providence, Rhode Island
  - Brown University, Providence, Rhode Island